CLINICAL TRIAL: NCT04879836
Title: Retrospective Analysis of the Effects of a Gum Gel Intended to Treat Signs and Symptoms of Teething in Infants
Brief Title: Effects of a Gum Gel Intended to Treat Signs and Symptoms of Teething
Status: Completed | Type: Observational
Sponsor: University of Urbino "Carlo Bo" (Other)
Responsible Party: Principal Investigator, Davide Sisti, PhD, University of Urbino "Carlo Bo"
Other Study IDs: UniUrb_GumGel_2021
Record Dates: First submitted 2021-05-04; First posted 2021-05-10 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Tooth Eruption Disorder
Keywords: gums; redness; fever; paediatric; inappetence; sleep disturbance
MeSH Terms: conditions — Erythema; Fever; Anorexia; Parasomnias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Teething Ring + Teething Gel
  Interventions: Device: Teething Gel; Device: Teething Ring
- Teething Ring
  Interventions: Device: Teething Ring

INTERVENTIONS:
Device: Teething Gel — Dosage: application of an even coat of 1mm thickness Frequency: 5 times/day (after main meals and before sleeping) Duration: 4 weeks
  Groups: Teething Ring + Teething Gel
Device: Teething Ring — The teething ring was filled with a coolant Usage: 5/10 min per time Frequency: 5 times/day Duration: 4 weeks

SUMMARY:
Teething discomfort is a widespread disorder affecting a very high percentage of infants. The use of hyaluronic acid gels has been shown in the last 20 years to be an effective tool, generally devoid of side effects, in reducing oral mucosal inflammation in adults. Its effectiveness in infants is affected by the strength of hyaluronic acid retention over the oral mucosa. This is in turn affected by formulation and may vary between different products due to the different ingredients used. In this study, the results collected by monitoring the paediatric experience regarding a newly developed HA-based medical device, intended to counteract teething discomfort in infants, will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Teething discomfort
* Being healthy (except for teething discomfort)

Exclusion Criteria:

* Being placed on one of the following therapies in the 45 days prior to the beginning of the study: immunosuppressive, cytotoxic, cortisone, antibiotics, antifungal and hormone therapy

Ages: 2 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants, without ethnic limitations, of both sexes and between the ages of 2 and 12 months, affected by teething discomfort but considered otherwise healthy.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Unexplained cry | 1 month (1 check per week)
  5-level Likert scale completed by the paediatrician
Irritability | 1 month (1 check per week)
  5-level Likert scale completed by the paediatrician
Sleep disturbance | 1 month (1 check per week)
  5-level Likert scale completed by the paediatrician
Inappetence | 1 month (1 check per week)
  5-level Likert scale completed by the paediatrician
Salivation | 1 month (1 check per week)
  5-level Likert scale completed by the paediatrician
Gum redness | 1 month (1 check per week)
  5-level Likert scale completed by the paediatrician
Fever | 1 month (1 check per week)
  Number of days with fever
General well-being | 1 month (1 check per week)
  5-level Likert scale completed by the paediatrician

CONTACTS AND LOCATIONS:
Overall Officials: Davide Sisti, PhD, Principal Investigator — University of Urbino "Carlo Bo"
Locations (1):
- University of Urbino Carlo Bo, Urbino, Italy